CLINICAL TRIAL: NCT06894654
Title: DERMATOMICS: Identifying Regulators of Skin Homeostasis
Acronym: DERMATOMICS
Status: Recruiting | Type: Observational
Sponsor: Relation Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: RRx-Profiling-002
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Systemic Sclerosis (SSc)
Keywords: Scleroderma; Skin; systemic sclerosis; SSc
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 10ml blood and skin samples collected from skin punch biopsies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Early SSc cohort: Early diagnosis of systemic sclerosis (SSc)
  Interventions: Procedure: Skin punch biopsy; Other: blood sampling; Behavioral: Questionnaire
- Late SSc cohort: Late diagnosis of systemic sclerosis (SSc)
  Interventions: Procedure: Skin punch biopsy; Other: blood sampling; Behavioral: Questionnaire
- Healthy cohort (control): Absence of SSc and Raynaud's Phenomenon (controls for the SSc cohorts)
  Interventions: Procedure: Skin punch biopsy; Other: blood sampling; Behavioral: Questionnaire

INTERVENTIONS:
Procedure: Skin punch biopsy — Skin punch biopsies are 5mm for this study. Participants with SSc will undergo 4 biopsies (2 in diseased area, 2 in non-diseased area if available). Healthy Volunteers will undergo 2 biopsies.
Other: blood sampling — 10mls blood will be taken for analysis and DNA sequencing
Behavioral: Questionnaire — All participants are required to complete a questionnaire with information on demographics, lifestyle, medical and medication history.

SUMMARY:
Diseases of the skin associated with chronic immune driven conditions, including scleroderma, lupus, dermatomyositis, psoriasis, and atopic dermatitis, significantly impact skin integrity, function, and overall quality of life. These conditions can lead to severe disfigurement, discomfort, and systemic complications, necessitating long-term medical intervention. The prevalence of these skin disorders is rising globally, driven by genetic, environmental, and immunological factors. Unravelling the mechanisms leading to skin manifestations may shed further insights in the overall mechanisms of disease.

The DERMATOMICS study will focus on understanding systemic sclerosis (SSc) biology.

Systemic Sclerosis (SSc) is a highly heterogeneous rare autoimmune fibrotic condition affecting the skin and internal organs. SSc is classified as a Connective Tissue Disease (CTD), a family of conditions including Systemic Lupus Erythematosus, Sjogren Syndrome and Inflammatory Myositis, all characterised by an autoimmune process affecting the connective tissue of most organs, communed by the presence of anti-nuclear antibodies (ANA). In SSc, patients are affected by a combination of tissue and vascular fibrosis, on the background of a chronic inflammatory process, leading to the highest per patient morbidity and mortality across CTDs. The main driver of mortality to date is interstitial lung disease (ILD), which is the consequence of the fibrotic involvement of the lungs, leading to a progressive loss of functional lung volumes, and ultimately, derangement of lung circulation, hypoxia, increased risk of hospitalisation for lower respiratory infections and death.

Current treatments for CTDs include general immunosuppressive treatments, not necessarily targeted to the specific mechanisms underlying their presentation, focusing on reducing inflammation and managing symptoms rather than addressing the underlying causes. Many of these therapies have limited effectiveness or are burdened with significant side effects. Therefore, there is a critical need to develop a comprehensive understanding of the cellular and molecular mechanisms underlying these disorders to identify novel therapeutic targets.

Several factors contribute to the risk and severity of SSc, including genetic predisposition, environmental triggers, immune system dysregulation, and lifestyle factors such as diet and smoking. The interactions between these factors are complex and not fully understood. By recruiting participants with SSc, we aim to obtain skin punch biopsies for detailed molecular and genetic analysis. To increase the informative value of our study we plan to implement an extreme phenotype approach and include participants with opposite degrees of severity.

Our study aims to elucidate the relationships between the molecular biology of skin cells, skin structure, genetic factors ("DNA"), and environmental influences. The goal is to identify and validate novel therapeutic targets that can lead to more effective and personalised treatment options for SSc, and more broadly for CTDs and CTD-associated skin and lung disease.

Modern single-cell technologies will be employed to dissect the cellular diversity within the skin. These advanced techniques have revolutionised our understanding of many tissues, but skin tissues remain underexplored, especially in the context of chronic skin diseases. Protocols for skin punch biopsy and single-cell profiling are well-established, allowing us to systematically analyse how genetic variations influence skin structure and function.

ELIGIBILITY:
Inclusion Criteria:

SSc participant cohort:

1. Age of 18 years inclusive, or older at the time of signing the informed consent
2. Documented diagnosis of systemic scleroderma (SSc) (early or late diagnosis)

Healthy cohort:

1. Approximate age/sex matching (majority of healthy participants to be recruited after cohort 1 and 2)
2. Absence of Raynaud's Phenomenon
3. Absence of lung disease
4. Not on immunosuppressive treatment

Exclusion Criteria:

SSc participant cohort:

1. Participants unable to provide informed consent.
2. Participants with suspected/established underlying malignancy.
3. Participants with suspected/established skin cancer.
4. Participants with suspected/established bloodborne disease.
5. Current enrolment or past participation in a study involving an investigational drug within 3 months or 5 half-lives of the investigational drug treatment (whichever is longer) before the day of sample collection.
6. Participants treated with cellular therapies, e.g., HSCT, Car-T cells, T cell engagers.
7. Participants treated with B-cell depletion therapies within 6 months.
8. Concurrent diagnosis of any other connective tissue disease (CTD) in overlap.
9. Diagnosis of other non-SSc dermatological conditions.
10. Systemic sclerosis-like illness, including but not limited to localised scleroderma (morphoea), eosinophilic fasciitis, sclerodermoid graft-versus-host disease, fibro mucinous conditions (scleredema, scleromyxedema), scleroderma-like conditions that are associated with environmental chemical and drug exposure (e.g., toxic rapeseed oil, vinyl chloride, bleomycin, gadolinium-based contrast agents [nephrogenic systemic fibrosis], or due to metabolic disease).
11. History or presence of significant non-sclereoderma related cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematologic, neurological disorders, or treatments for those, capable of significantly interfering with the results and interpretation of data.
12. Smoking history (5 years smoke free acceptable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with either early systemic sclerosis (SSc) or late systemic sclerosis (SSc)
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2030-11-01 (Estimated)

PRIMARY OUTCOMES:
Acquisition of skin samples | Within 48 hours of sampling
  Skin samples acquired from skin punch biopsies to be used for the study of RNA.

SECONDARY OUTCOMES:
Acquisition of 10ml of blood | Within 48 hours of sampling
  Blood to use used for genetic sequencing, and/or other downstream omics/assays
Completion of participant questionnaire | EDC entry within 1 week of skin & blood samples being taken.
  Participant metadata to be used to understand cohort and identify confounding factors

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Chapel Allerton Hospital, Leeds
  - Royal Free Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
A pharmaceutical partner is providing funding support to a research collaboration with Relation Therapeutics and will be involved in data review.
  It is intended that the results of the study will be published when appropriate. There will be no reference in the study results / reports / publications to any information that would identify participants. The final dataset, which may include a small number of select fields from the EDC database, will not contain any identifiable personal data.
Time Frame: Data will not be released until the study is complete. Raw data files in the original format (e.g. fastq) and the accompanying anonymised phenotypic data will be uploaded to a public repository e.g. the NCBI database of Genotypes and Phenotypes (dbGaP) at https://www.ncbi.nlm.nih.gov/gap/.
Access Criteria: Any database selected to host genetic data must require legally-binding data access agreements with participating researchers.